CLINICAL TRIAL: NCT04984434
Title: A First-in-human, Open-label, Multiple Center Phase 1 Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetic, Immunogenicity, and Preliminary Efficacy of F182112 in Patients With Relapsed or Refractory Multiple Myeloma.
Brief Title: Phase 1 Study of F182112 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F182112-001
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Dose-Escalation Study, Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single Arm (Experimental)
  Interventions: Drug: F182112

INTERVENTIONS:
Drug: F182112 — Eight dose cohorts: 0.01, 0.1, 0.3, 1, 3, 10, 20 and 30 μg/kg) d1 treat every weeks.

SUMMARY:
This trial is a Multiple center, Open-label, dose escalation Phase Ⅰ clinical study. The purpose is to evaluate the safety and tolerability of F182112 when infused intravenously (IV) and determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of F182112 when infused IV.

DETAILED DESCRIPTION:
To assess the safety, tolerability, and dose-limiting toxicities (DLTs) and to determine a recommended phase 2 dose regimen (RP2DR) of F182112 as monotherapy in patients with relapsed or refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* 1) Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures;

  2) Male or female ≥ 18 years;

  3) Patient has a history of multiple myeloma with relapsed and refractory disease, and must:
  1. Relapsed after an autologous stem cell transplant (ASCT), or not suitable for ASCT;
  2. Must have received at least 2 prior multiple myeloma treatment regimens (not including autologous stem cell transplant) including a proteasome inhibitor, an immunomodulatory agent;

     4) ECOG of 0-2;

     5) Patients must have measurable disease, including at least one of the criteria below:

  <!-- -->

  1. M-protein ≥ 0.5 g/dL by SPEP/immunofixation or
  2. ≥ 200 mg/24 hours urine collection by UPEP or
  3. Serum free light chain (FLC) levels > 100 mg/L (milligrams/liter involved light chain) and an abnormal kappa/lambda (κ/λ) ratio in patients without detectable serum or urine M-protein;

     6) Adequate hepatic function as evidenced by meeting all the following requirements:

  <!-- -->

  1. Blood routine: absolute neutrophil count (ANC) ≥ 1.0×109/L, hemoglobin (Hb) ≥70g/L, Platelet ≥ 50×109/L;
  2. Liver function: total bilirubin ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 2.5 × ULN, Aspartate aminotransferase (AST) ≤ 2.5 × ULN;
  3. Renal function: calculated creatinine clearance (CrCL) ≥ 30 mL/min (Cockroft-Gault Equation).

     7) Recovery to Grade 0-1 from adverse events related to prior anticancer therapy except alopecia, ≤ Grade 2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy.

     Exclusion Criteria:
* 1) Patient has primary light chain amyloidosis or plasma cell leukemia;

  2) Patient has symptomatic central nervous system involvement of multiple myeloma;

  3) Received systemic anti-myeloma therapy within 2 weeks, or received plasma exchange within 4 weeks;

  4) Received any experimental drugs within 4 weeks or 5 half-lives (whichever is shorter);

  5) Patient has received ≥ 40 mg/day dexamethasone equivalent within 7 days before starting F182112. Short term use of corticosteroids at doses equivalent to > 10 mg/d of prednisone；

  6) Received any monoclonal antibody therapy within 30 days;

  7) Prior treatment with any B cell maturation antigen (BCMA) targeted therapy;

  8) Patient had a prior allogeneic stem cell transplant or had a prior autologous stem cell transplant ≤ 3 months prior to starting F182112;

  9) Live virus vaccine within 30 days prior to study entry;

  10) Major surgery within 4 weeks prior to study entry;

  11) Concurrent malignancy within 3 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer under active surveillance, prostate cancer that has undergone definitive treatment, ductal carcinoma in situ of the breast, or ≤ T1 urothelial carcinoma;

  12) Patients with active mucosa or visceral bleeding;

  13) Severe cardiovascular disease, including CVA, TIA, myocardial infarction, or unstable angina within 6 months of study entry; NYHA class III or IV heart failure within 6 months of study entry; Uncontrolled arrhythmia within 6 months of study entry. Patients with a rate-controlled arrhythmia may be eligible for study entry at the discretion of the Medical Monitor;

  14) Active infection requiring antibiotic, antiviral or antifungul therapy;

  15) Active viral hepatitis;

  16) Has a history of immunodeficiency, include HIV infection;

  17) Treponema pallidum infection;

  18) Received any experimental drugs or anti-tumor drugs within 2 weeks;

  19) Subject has any condition that confounds the ability to interpret data from the study;

  20) Females and males must practice true abstinence or agree to contraceptive methods throughout the study, and 6 months after the last giving F182112;

  21) Any condition that the investigator or primary physician believes may not be appropriate for participating the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
DLTs | Up to 28 days
  Incidence of dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period
Maximum Tolerated Dose (MTD) | Approximately 12 months
  Maximum Tolerated Dose
RP2D | Approximately 12 months
  Preliminary Antitumor Activity of F182112 at the RP2D(s) in Part 2

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 24 months
  To evaluate the duration from the first dose to death of patients with MM for any reason.
Progression-free survival (PFS) | Approximately 24 months
  Evaluation of the efficacy of F182112 in patients with MM on progression-free survival.
Objective response rate (ORR) | Approximately 24 months
  Objective remission rate was used to evaluate the efficacy of F182112 injection in patients with MM.

OTHER OUTCOMES:
Minimal Residual Disease (MRD) Negative Rate | Approximately 24 months
  Minimal Residual Disease (MRD) Negative Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shaohong Yin, Linyi, Shandong, China